CLINICAL TRIAL: NCT07354659
Title: A Randomized, Blinded, Placebo- and Active-Controlled, Adaptive Phase 2 Study to Evaluate the Immunogenicity and Safety of SYS6017 (a Herpes Zoster mRNA Vaccine) in Healthy Participants Aged 40 Years and Above
Brief Title: Immunogenicity and Safety of SYS6017 in the Participants Aged 40 Years and Above
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SYS6017-002
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Randomized, placebo or active-controlled, Masking
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dosage A of zoster mRNA vaccine SYS6017 (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Dosage B of zoster mRNA vaccine SYS6017 (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Dosage C of zoster mRNA vaccine SYS6017 (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Dosage D of zoster mRNA vaccine SYS6017 (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Dosage E of zoster mRNA vaccine SYS6017 (Experimental)
  Interventions: Biological: A zoster mRNA vaccine SYS6017
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Active Comparator Vaccine (Active Comparator)
  Interventions: Biological: Active Comparator Vaccine

INTERVENTIONS:
Biological: A zoster mRNA vaccine SYS6017 — SYS6017，two-dose vaccination schedule (Month 0, 2)
  Arms: Dosage A of zoster mRNA vaccine SYS6017; Dosage B of zoster mRNA vaccine SYS6017; Dosage C of zoster mRNA vaccine SYS6017; Dosage D of zoster mRNA vaccine SYS6017; Dosage E of zoster mRNA vaccine SYS6017
Other: Placebo — 0.9% saline，two-dose vaccination schedule (Month 0, 2)
  Arms: Placebo
Biological: Active Comparator Vaccine — Recombinant Zoster Vaccine (CHO cell)，two-dose vaccination schedule (Month 0, 2)
  Arms: Active Comparator Vaccine

SUMMARY:
Herpes zoster is caused by the reactivation of latent varicella-zoster virus (VZV) which stays in latency after its primary infection. Immunosenescence contributes significantly to elevating morbidity associated with aging. Vaccination plays a key role in reducing the disease burden of zoster and the associated complications. We are conducting a study entitled "A Randomized, Blinded, Placebo- and Active-Controlled, Adaptive Phase 2 Clinical Trial to Evaluate the Immunogenicity and Safety of SYS6017 (a Herpes Zoster mRNA Vaccine) in Healthy Participants Aged 40 Years and Above".

ELIGIBILITY:
Inclusion Criteria:

* 1. Individuals aged 40 years or older;
* 2. Able to understand the study procedures, comply with the protocol requirements to attend all the scheduled visits, voluntarily consent to participate in the study, and sign the informed consent form;
* 3. Is physically eligible at the discretion of investigators based on medical history inquiry and physical examination; For participants with chronic underlying diseases (e.g., diabetes mellitus, hypertension, hyperlipidemia and other chronic conditions), they may be enrolled if their conditions have been well controlled within 3 months prior to enrollment in this study (i.e., additional medical interventions or major adjustments to treatments are not required);
* 4. For female participants of childbearing potential: No sexual activity or effective contraceptive methods were used within one menstrual cycle before enrollment; No pregnancy plans and agree to adopt effective contraceptive methods within 8 months after enrollment.

Exclusion Criteria:

* 1. History of zoster;
* 2. History of vaccination with varicella vaccine or zoster vaccine (including investigational vaccine);
* 3. Axillary temperature ≥ 37.1℃ on the day of enrollment or within 24 h before enrollment;
* 4. History of allergy to any component of the investigational vaccine; or history of severe allergic reactions to vaccines or medications (including but not limited to anaphylaxis, allergic laryngeal edema, Henoch-Schönlein purpura, thrombocytopenic purpura, or Arthus reaction);
* 5. History of myocarditis, pericarditis, or idiopathic cardiomyopathy, or any condition that could increases the risk of myocarditis or pericarditis
* 6. History of demyelinating diseases, including but not limited to Guillain-Barré syndrome, multiple sclerosis, ophthalmoneuromyelitis, acute disseminated encephalomyelitis, etc.;
* 7. Current epilepsy or convulsion, severe neurological or psychiatric disorders;
* 8. Have contraindications to intramuscular injection, e.g., diagnosed thrombocytopenia, any coagulation disorders, or ongoing treatment with anticoagulants, etc.;
* 9. Active malignant tumor, malignant tumor without adequate treatment, malignant tumor with a potential risk of recurrence during the study;
* 10. Active, unstable, severe or uncontrolled cardiovascular and cerebrovascular diseases, thrombotic diseases, blood and lymphatic system diseases, liver and kidney diseases, respiratory diseases, metabolic diseases, musculoskeletal diseases, autoimmune diseases, etc;
* 11. History of diagnosed immunocompromise or immunosuppression, congenital or functional asplenia, or splenectomy before enrollment;
* 12. Long-term (defined as more than 14 consecutive days) systemic use of immunosuppressants, immunostimulants, or other immunomodulatory drugs (e.g., corticosteroids at a dose of ≥ 20 mg/day prednisone or equivalent) within 6 months prior to enrollment; however, inhaled and topical corticosteroids are permitted; or planned administration of the aforementioned agents during the study period;
* 13. Administration of whole blood, plasma, serum, immunoglobulin, or monoclonal antibodies within 3 months prior to enrollment, or planned administration of the aforementioned products during the study period;
* 14. Blood donation or blood loss ≥ 450 mL within one month before enrollment, or planning to donate blood during the study;
* 15. Vaccination with any other vaccines within 30 days prior to enrollment, or planned vaccination with any other vaccines within 30 days after the last dose of the study vaccine;
* 16. Current participation in or planned participation in other clinical trials during the study period;
* 17. For female participants of childbearing potential: positive pregnancy test result prior to enrollment, current pregnancy or lactation, or planned pregnancy within 8 months after enrollment;
* 18. Unable to comply with the study procedures and requirements, or presence of other conditions that make the participant inappropriate for this clinical trial, as judged by the investigators.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
solicited adverse events | within 14 days post each vaccination
unsolicited adverse events | within 30 days post each vaccination
Geometric Mean Concentration (GMC) of anti-gE antibody | On Day 14 and Day 30 after the completion of the full vaccination course
Geometric Mean Fold Increase (GMFI) of anti-gE antibody | On Day 14 and Day 30 after the completion of the full vaccination course
Seroconversion Rate (SCR) of anti-gE antibody | On Day 14 and Day 30 after the completion of the full vaccination course

SECONDARY OUTCOMES:
serious adverse events | from the first vaccination through 12 months post the second vaccination
adverse events of special interest | from the first vaccination through 12 months post the second vaccination
pregnancy events reported by the participants | from the first vaccination through 12 months post the second vaccination
Geometric Mean Titer (GMT) of anti-VZV antibody | On Day 14 after the completion of the full vaccination course
Geometric Mean Fold Increase (GMFI) of anti-VZV antibody | On Day 14 after the completion of the full vaccination course
Seroconversion Rate (SCR) of anti-VZV antibody | On Day 14 after the completion of the full vaccination course
cellular immune response | On Day 14 and Day 30 after the completion of the full vaccination course
  the frequency of peripheral blood mononuclear cell (PBMC) secreting gE-specific cytokines